CLINICAL TRIAL: NCT03682458
Title: Study of Neurological Pathological Mechanisms of and Neurodegenerative Diseases in Neurons and Glia Derived From Induced Stem Cells (iPS) in Patients and Healthy Family Controls.
Brief Title: Study of Neurodegenerative Diseases Induced Stem Cells in Patients and Healthy Family Controls.
Acronym: NeuronsiPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Collaborators: San Raffaele University Hospital, Italy (Other)
Responsible Party: Principal Investigator, Stefano Gambardella, Principal Investigator, Neuromed IRCCS
Other Study IDs: CGM-02
Record Dates: First submitted 2018-09-17; First posted 2018-09-24 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Neurodegenerative Diseases
Keywords: iPS; genetic mutations; neurodegenerative diseases; experimental therapeutic approaches; molecular processes
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Study of Neurodegenerative Diseases Induced Stem Cells — The aim of this study is to generate iPS-induced stem cell lines from patients with neurological and neurodegenerative diseases to differentiate into neurons and glial cells to study the pathological cellular and molecular processes of these diseases. These in vitro cultures will also be used to validate molecules or experimental therapeutic approaches. IPS cells will be generated by the reprogramming of isolated 10-mL cells of peripheral venous blood.

SUMMARY:
Neurological and neurodegenerative diseases have a major impact in families and in the national health service due to the lack in many cases of effective and long-lasting therapies. The lack of these therapeutic strategies is due in large part to the difficulty of modeling these pathologies in vitro. In fact, the impossibility of being able to cultivate human neurons in vitro has forced the use of animal cell models that do not adequately recapitulate the complexity of these human pathologies. For this reason it is necessary to proceed with the development of in vitro models of human origin that reproduce the molecular and biochemical characteristics of these diseases.

The discovery of cellular reprogramming allowed the generation of pluripotent stem cells from the conversion of somatic cells taken from adult individuals.

The proposing group already has great experience in generating iPS cells by reprogramming and in differentiating them into neurons and glias useful for neurological disease cellular studies. As an example, Dr. Broccoli's group has generated iPS cells from patients with Parkinson's disease and mutations in the OPA1 gene. The study of neurons differentiated by these iPS cells allowed to identify mitochondrial defects at the base of neuronal dysfunctions and to identify for the first time how the degeneration of dopaminergic neurons also depends on a moving mode of cell death called necroptosis.

The investigators therefore propose to establish lines of iPS cells from patients with genetic mutations responsible for neurological and neurodegenerative diseases to generate neuronal and glial models in vitro for the study of pathological mechanisms and the validation of new future experimental therapies.

DETAILED DESCRIPTION:
1. INTRODUCTION Neurological and neurodegenerative diseases have a major impact in families and in the national health service due to the lack in many cases of effective and long-lasting therapies. The lack of these therapeutic strategies is due in large part to the difficulty of modeling these pathologies in vitro. In fact, the impossibility of being able to cultivate human neurons in vitro has forced the use of animal cell models that do not adequately recapitulate the complexity of these human pathologies. For this reason it is necessary to proceed with the development of in vitro models of human origin that reproduce the molecular and biochemical characteristics of these diseases.

   The discovery of cellular reprogramming allowed the generation of pluripotent stem cells from the conversion of somatic cells taken from adult individuals. This technology is based on the expression of the 4 genes OCT4, SOX2, KLF4 and c-MYC that synergistically are sufficient to convert somatic cells into induced stem cells called iPS (1,2). For this technology Prof. S. Yamanaka from the University of Kyoto was awarded the Nobel Prize for Medicine in 2012 (3). Human iPS-induced stem cells can be maintained in vitro in a stable manner over time and then be differentiated into any specialized cell including neurons and glial cells. In this way, therefore, it is possible to generate human neurons from adult individuals suffering from neurological pathologies, allowing the study of pathophysiological mechanisms in cells affected by these diseases. Research in recent years has established many reliable protocols to differentiate human iPS cells into different subtypes of neurons (glutamatergics, GABAergics, dopaminergics), astrocytes, oligodendrocytes and microglia (4-6). Thanks to these procedures it was possible to generate neuronal and glial models of many neurological diseases by creating very useful systems for studying pathological processes and identifying new therapeutic targets for some genetic forms of Alzheimer's, Parkinson's and autism (7-9).

   The proposing group already has great experience in generating iPS cells by reprogramming and in differentiating them into neurons and glias useful for neurological disease cellular studies. As an example, Dr. Broccoli's group has generated iPS cells from patients with Parkinson's disease and mutations in the OPA1 gene (8). The study of neurons differentiated by these iPS cells allowed to identify mitochondrial defects at the base of neuronal dysfunctions and to identify for the first time how the degeneration of dopaminergic neurons also depends on a moving mode of cell death called necroptosis (8).

   The investigators therefore propose to establish lines of iPS cells from patients with genetic mutations responsible for neurological and neurodegenerative diseases to generate neuronal and glial models in vitro for the study of pathological mechanisms and the validation of new future experimental therapies.
2. PURPOSE AND DRAWING OF THE STUDY The aim of this study is to generate iPS-induced stem cell lines from patients with neurological and neurodegenerative diseases to differentiate into neurons and glial cells to study the pathological cellular and molecular processes of these diseases. These in vitro cultures will also be used to validate molecules or experimental therapeutic approaches. IPS cells will be generated by the reprogramming of isolated 10-mL cells of peripheral venous blood.

The study therefore involves taking 10 ml of peripheral blood from

1. Subjects carrying genetic mutations that condition the development of neurological and / or neurodegenerative diseases.
2. Relatives or family control non-carriers of genetic mutations conditioning the development of metabolic and / or neurodegenerative diseases (healthy donors).

3. EXPERIMENTAL PHASE

1. Following a Neurological visit, a Neurological Consultation is requested by the Neurologist.
2. Genetic Counseling is performed and the molecular test to be performed is identified. Classical diagnostic paths are applied according to specific national guidelines for each pathology (SIGU: http://www.sigu.net/show/attivita/5/1/LINEE%20GUIDA%20SIGU) that indicate the analysis of the most suitable to analyze and above all more frequently involved.
3. A blood sample is taken after signing an informed consent form (informed consent Neuromed version 12.02.2015) for the diagnostic study. Approximately 10 milliliters of blood will be taken and subsequently a part will be fractionated in serum and lymphocytes which will be stored at -80 ° C.
4. Molecular analyzes are carried out at the Center for Molecular Genetics of the IRCCS INM Neuromed Institute through NGS or Sanger Sequencing, Multiplex Ligation-dependent Probe Amplification (MLPA) and Microsatellites.
5. If the molecular diagnosis has identified a gene and / or a variant of interest compatible with the clinical phenotype, or has identified a variant with uncertain clinical significance (VoUS), the real scientific importance of generating the patient's iPS stem cells is evaluated in object
6. If the possibility of generating such cells is positively evaluated, during consultation, at the same time as the withdrawal of the report, the patient is asked for his consent (informed consent Neuromed version 12.02.2015) to participate in this research protocol. A peripheral blood sample of 10 ml is performed.
7. Blood samples in tubes with EDTA as anticoagulant are sent by express courier to the laboratory of Dr. Vania Broccoli at the San Raffaele Hospital (OSR) where the mononuclear cells of the blood will be reprogrammed in iPS stem cells.
8. Part of the iPS stem cells generated in OSR will be sent to the NEUROMED to confirm the pathological mutation and the correct cell genetic
9. iPS stem cells will be differentiated into neurons and glia for the study of the pathological mechanisms underlying neuropathology.
10. iPS stem cell aliquots will be cryopreserved in liquid nitrogen both in OSR and in NEUROMED to ensure the maintenance of the lines that will be maintained until the end of the study.

4. MATERIALS AND METHODS Reprogramming of peripheral blood mononuclear cells Once the 10 ml of peripheral venous blood is obtained, mononuclear cells (PBMCs) will be isolated and reprogrammed using the Sendai RNA virus, which expresses the 4 genes SOX2, OCT4, KLF4 and c-MYC without integrating in the cell genome. This operation will be performed in sterile BL2 rooms available at the laboratory of Dr. Vania Broccoli at the Neuroscience Division of the San Raffaele Hospital in Milan.

Then the PBMCs will be then plated on a fibroblast mat in sterile 10 mm Petri dishes with a culture medium enriched with the cytokine bFGF (4ng / ml) (8). In these culture conditions, the first iPS reprogrammed stem cell clones will be visible after approximately 30 days. At this point, the individual clones will be isolated and grown to amplify the number of cells and establish proliferating lines. The progeny of the single clones will be studied to verify the correct reprogramming in pluripotent stem cells through: 1) activation of marker genes of the state of pluripotent staminality (Nanog, Sox2, Oct4, SEEA4), capacity of in vitro differentiation in the somatic cells of the three sheets embryonic endoderm, mesoderm and ectoderm, minimal contamination of differentiated cells in the culture. Once the induced pluripotent stem cell generation (iPS) has been validated, the cells will be used to be differentiated into different neuronal and glial types for experiments aimed at understanding and describing the pathogenetic mechanisms of the subject's study diseases. For the generation of neurons will be followed the protocol developed by Shi and colleagues (5) that uses retinoic acid and TGFbeta / BMP proteins inhibitors to direct the neuroectodermal differentiation. This procedure has already been validated and used in our laboratories demonstrating the differentiation of iPS stem cells into mature and functioning neurons (10) (Figure 1).

Once the processes of differentiation with iPS stem cells have been established, the investigators will proceed with the analysis of the phenotype in the patients' cells with respect to controls derived from healthy controls. In particular, with regard to the analyzes in neurons, survival parameters will be investigated, neuronal activity through electrophysiological recordings, mitochondrial morphology and metabolism, endoplasmic reticulum stress, and synapse formation and functioning. For glial cells the levels of inflammation including the activity of TNF-alpha, IL-1beta, IL-4, IL-6 and NOS proteins will be analyzed. Along with these studies, a genomic analysis will be carried out by comparing the gene expression profiles of neurons and glial cells. The analysis will be done for RNA-Seq, a "next-generation sequencing" technique that allows to analyze the expression levels of all genes in the genome. The genes thus identified will be validated with real-time PCR analysis and their functioning will be investigated in neurons and cells derived from the patient's cells.

5. STATISTICS For the study of pathological processes 6 lines of iPS cells will be derived from each patient and healthy individual. The investigators anticipate from our previous experience that the comparison between this number of lines between patient and healthy donor is more than sufficient to have statistical significance for the different in vitro experiments that will be performed. In case it will be possible to generate new lines of iPS cells from the same patient in the unlikely event it was necessary.

6. ETHICAL ASPECTS The procedures reported in the study concerning conducting, conducting and documentation are designed to ensure that the ethical principles set forth in the Helsinki Declaration and its revisions are upheld. The study will be conducted taking into account regulatory requirements and legal obligations. In particular, the normative reference is represented by the DL n.211, 24/06/2003 and DM 17/12/2004 on non-profit studies. Furthermore, before enrollment, all potentially eligible patients will receive complete and comprehensive information on the study. In order to be enrolled it will be necessary that the patients consent to the participation in the study and processing of personal data, according to the law 196/03 on the protection of persons and the processing of personal data. The informed consent previously approved by the ethics committee will be used.

7. FINAL OBJECTIVES This program aims to identify the sub-cellular processes altered exactly in human cells (neurons and i) affected by the neuropathologies in question. Furthermore, this study will also allow us to integrate molecular data with the aim of identifying genes whose specific alterations may underlie these cellular dysfunctions. The ultimate aim of this experimental program is to identify the alteration of specific molecular mechanisms underlying these diseases. These new knowledge will be essential to think about the development of new translational strategies based on pharmacological approaches or gene therapy. This is of great importance since the diseases in question are orphans of effective treatment and limited to exclusively symptomatic treatments.

8. PROJECT COSTS Molecular diagnostics is performed routinely at the Molecular Genetics Center of IRCCS Neuromed. There are no additional costs as the analyzes are part of diagnostic procedures carried out in agreement with the NHS.

IPS generation is performed by IRCCS San Raffaele. The costs for the development of these lines are therefore completely dependent on them.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of neurodegenerative disease
* identification of gene variant of interest compatible with the clinical phenotype.

Exclusion Criteria:

* no identification of gene variant of interest compatible with the clinical phenotype.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Following a Neurological visit a Genetic Counseling is performed and the molecular test to be performed is identified.
  A blood sample is taken after signing an informed consent form (informed consent Neuromed version 12.02.2015) for the diagnostic study. The Molecular analyzes are carried out and If the molecular diagnosis has identified a gene and / or a variant of interest compatible with the clinical phenotype the mononuclear cells of the blood will be reprogrammed in iPS stem cells.
  iPS stem cells will be differentiated into neurons and glia for the study of the pathological mechanisms underlying neuropathology.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Study of Neurodegenerative Diseases Induced Stem Cells (iPS) in Patients and Healthy Family Controls. | 10 days
  1.Neurology consulting Clinical valuation

SECONDARY OUTCOMES:
Study of Neurodegenerative Diseases Induced Stem Cells (iPS) in Patients and Healthy Family Controls. | 1 day
  2. Genetic Counseling family history

OTHER OUTCOMES:
Study of Neurodegenerative Diseases Induced Stem Cells (iPS) in Patients and Healthy Family Controls. | 2 years
  3. Molecular testing
  * Molecular analysis
  * iPS stem cells will be differentiated into neurons and glia for the study of the pathological mechanisms underlying neuropathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Stefano Gambardella, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No